CLINICAL TRIAL: NCT06021015
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial on the Safety and Efficacy of Polyvinyl Alcohol Sodium Acrylate Embolization Microspheres for Transcatheter Arterial Chemoembolization of Colorectal Cancer Liver Metastases
Brief Title: Safety and Efficacy of Polyvinyl Alcohol Sodium Acrylate Embolization Microspheres for CRLM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEBIRI-TACE
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer Liver Metastasis
Keywords: colorectal cancer; liver metastasis; embolization microspheres; efficacy; safety; transcatheter arterial chemoembolization
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Irinotecan and polyvinyl alcohol sodium acrylate embolization microspheres（Unipearls®）
  Interventions: Device: Irinotecan and polyvinyl alcohol sodium acrylate embolization microspheres（Unipearls®）
- Control group (Active Comparator): Irinotecan and HepaSphere Microspheres
  Interventions: Device: Irinotecan and HepaSphere Microspheres

INTERVENTIONS:
Device: Irinotecan and polyvinyl alcohol sodium acrylate embolization microspheres（Unipearls®） — Irinotecan and polyvinyl alcohol sodium acrylate embolization microspheres（Unipearls®）
  Arms: Experimental group
Device: Irinotecan and HepaSphere Microspheres — Irinotecan and HepaSphere Microspheres
  Arms: Control group

SUMMARY:
This study is a prospective, multicenter, randomized controlled clinical trial to evaluate the safety and efficacy of polyvinyl alcohol sodium acrylate embolization microspheres and HepaSphere Microspheres loaded with irinotecan for the treatment of colorectal cancer with hepatic metastases through arterial chemoembolization.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled clinical trial. Seventy-two patients with colorectal cancer liver metastases that are not feasible or suitable for surgical resection will be enrolled in this study. The experimental group received transcatheter arterial chemoembolization (TACE) treatment with polyvinyl alcohol sodium acrylate embolization microspheres loaded with 100mg irinotecan and the control group received TACE treatment with HepaSphere Microspheres loaded with 100mg irinotecan. All patients received 1-2 TACE treatment as needed. The primary end point of this study is disease control rate (DCR) of target lesions 1 month after the last TACE treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 80 years old (including threshold), regardless of gender；
2. Imaging or pathology/cytology clearly diagnosed as colorectal cancer liver metastases, with complete resection of the primary lesion and no local recurrence;
3. Researchers believe that liver metastases are not feasible or suitable, or patients refuse surgical resection；
4. ECOG score ≤ 2 points, Child Pugh grade A or B；
5. At least one measurable liver metastasis with a diameter greater than 1 cm without embolization treatment (the maximum diameter of the target lesion is less than 10 cm)；
6. Voluntarily participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Patients with known severe allergy to contrast agents (iodine contrast agents, gadolinium contrast agents, etc.) or embolic materials (polyvinyl alcohol sodium acrylate copolymer) ;
2. White blood cell count<3.0×109/L, platelet count<75×109/L，hemoglobin<70 g/L；
3. Total bilirubin>2 times the upper limit of normal value, Alanine transaminase (ALT) or aspartate aminotransferase (AST) >5 times the upper limit of normal value, Alkaline phosphatase>2.5 times the upper limit of normal value, albumin<30 g/L;
4. Creatinine>1.5 times the upper limit of normal value, creatinine clearance rate<30 mL/min;
5. Prothrombin time and activated partial thromboplastin time>1.5 times the upper limit of normal value;
6. Target lesion blood supply artery cannot undergo TACE treatment (the blood supply artery is too thin，vasospasm or suspected vasospasm，peripheral vascular resistance of the blood supply artery hinders the entry of embolic microspheres into the lesion site，severe Atherosclerosis, etc) or there is a risk of embolism (collateral vascular pathway endangers normal areas, etc)；
7. The expected survival time is less than 3 months;
8. Patients who have received embolization therapy for the target lesion or undergo the first TACE treatment for the target lesion after enrollment and require combined ablation/radiotherapy;
9. Pregnant and lactating women, or those who plan to conceive during the study period;
10. Those who have participated in other intervention clinical trials within one month before the trial;
11. The researchers believe that the subjects are intolerant and other unsuitable candidates for participating in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) of target lesions 1 month after the last TACE treatment | 3 month
  Disease control rate (DCR) of target lesions 1 month after the last TACE treatment

SECONDARY OUTCOMES:
Success rate | 3 month
  The success rate of embolization techniques for target lesions
Disease control rate (DCR) of target lesions 1 month after first TACE treatment | 1 month
  Disease control rate (DCR) of target lesions 1 month after first TACE treatment
Objective response rate (ORR) | 3 month
  Objective response rate (ORR) of target lesions 1 month after the first TACE treatment and 1 month after the last TACE treatment
Equipment performance evaluation | 3 month
  Equipment performance evaluation: evaluation of conveying performance and degree of embolism

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital

IPD SHARING:
Plan to Share IPD: No